CLINICAL TRIAL: NCT02296580
Title: A Feasibility Study of the Nativis Voyager® System in Patients With Recurrent Glioblastoma Multiforme (GBM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nativis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAT-101
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Nativis Voyager RFE Therapy (Experimental): Subjects will be treated with Nativis Voyager therapy until tumor progression.
  Interventions: Device: Nativis Voyager RFE Therapy

INTERVENTIONS:
Device: Nativis Voyager RFE Therapy — Nativis Voyager Radiofrequency Energy Therapy

SUMMARY:
This feasibility study will assess the effects of the Nativis Voyager therapy in patients with first or second recurrence of GBM who have either failed standard of care or are intolerant to therapy. The study will enroll and treat up to 32 subjects with Voyager plus lomustine with or without bevacizumab. Safety and clinical utility will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subject has histologically confirmed diagnosis of GBM.
* Subject has failed or intolerant to radiotherapy.
* Subjects has failed or intolerant to temozolomide therapy.
* Subject has progressive disease with at least one measureable lesion on MRI.
* Subject is at least 18 years of age.
* Subject has a KPS ≥ 60.
* Subject has adequate organ and marrow function.

Exclusion Criteria:

* Subject has received bevacizumab (Avastin).
* Subjecting has any condition, including compromised pulmonary function, that would preclude the use of lomustine.
* Subject is currently being treated with other investigational agents.
* Subject has received other investigational therapy within the last 28 days.
* Subject has received surgery within the last four weeks.
* Subject is within 12 weeks of completion of radiation.
* Subject has an active implantable or other electromagnetic device.
* Subject has a metal implant, including a programmable shunt, in the head or neck that is incompatible with MRI.
* Subject is known to be HIV positive.
* Subject is pregnant, nursing or intends to become pregnant during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Number of any adverse events associated with the investigational therapy. | Through one month following investigational treatment
  Safety Assessment as assessed by adverse events

SECONDARY OUTCOMES:
Clinical Utility: PFS | Six months
  Progression Free Survival as assessed by RANO
Clinical Utility: OS | 18 months
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Donna Morgan Murray, PhD, Study Director — Nativis, Inc.
Locations (13):
- United States (12):
  - University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Center for Neurosciences, Tucson, Arizona
  - cCARE - California Cancer Associates for Research & Excellence, Encinitas, California
  - John Wayne Cancer Institute @ Providecne St. Johns Health Center, Santa Monica, California
  - Associated Neurologists of Southern CT, P.C., Fairfield, Connecticut
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - University of Kansas Medical Center (KUMC), Kansas City, Kansas
  - Providence Brain & Spine Institute, Portland, Oregon
  - Cancer Care Collaborative, Austin, Texas
  - Baylor Scott & White Health, Temple, Texas
  - Virginia Mason Hospital & Medical Center, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
- St Vincent's Hospital Melbourne, Melbourne, Australia

REFERENCES:
- [Derived] Barkhoudarian G, Badruddoja M, Blondin N, Chowdhary S, Cobbs C, Duic JP, Flores JP, Fonkem E, McClay E, Nabors LB, Salacz M, Taylor L, Vaillant B, Gill J, Kesari S. An expanded safety/feasibility study of the EMulate Therapeutics Voyager System in patients with recurrent glioblastoma. CNS Oncol. 2023 Sep 1;12(3):CNS102. doi: 10.2217/cns-2022-0016. Epub 2023 Jul 18. PMID 37462385